CLINICAL TRIAL: NCT02699515
Title: A Phase I, Open-label, Multiple-ascending Dose Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Biological and Clinical Activity of MSB0011359C (M7824) in Subjects With Metastatic or Locally Advanced Solid Tumors With Expansion to Selected Indications in Asia
Brief Title: MSB0011359C (M7824) in Participants With Metastatic or Locally Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200647-0008
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumors
Keywords: MSB0011359C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSB0011359C (M7824) (Experimental)
  Interventions: Drug: MSB0011359C

INTERVENTIONS:
Drug: MSB0011359C — Subjects with metastatic or locally advanced solid tumors received intravenous infusion of MSB0011359C over 1 hour once every two weeks for up to 12 months until confirmed progressive disease (PD), unacceptable toxicity, or any criterion for withdrawal from the trial or investigational medicinal product (IMP) occurs.
  Other Names: M7824

SUMMARY:
The main purpose of this study was to assess the safety and tolerability of MSB0011359C. Study consists of dose-escalation part and an expansion part in participants with metastatic or locally advanced solid tumors, for which no standard effective therapy exists or a standard therapy had failed.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent and had signed the appropriate written informed consent form (ICF), prior to performance of any trial activities
* Eligible male and female participants aged greater than or equal to (>=)20 years
* Histologically or cytologically proven metastatic or locally advanced solid tumors, for which no effective standard therapy exists or standard therapy had failed
* Eastern Cooperative Oncology Group performance status (ECOG) performance status of 0 to 1 at trial entry
* Life expectancy >=12 weeks as judged by the Investigator.
* Adequate hematological function defined by white blood cell (WBC) count >=3*10^9/Liter with absolute neutrophil count (ANC) >=1.5*10^9/Liter, lymphocyte count >=0.5* 10^9/Liter, platelet count >=75*10^9/Liter, and Hemoglobin (Hgb) >= 9 grams per deciliter (g/dL) (in absence of blood transfusion)
* Adequate hepatic function defined by a total bilirubin level <=1.5 × Upper limit of normal (ULN), an AST level <= 2.5 × ULN, and an ALT level <= 2.5 × ULN
* Adequate renal function defined by an estimated creatinine clearance >50 milliliter per minute (mL/min) according to the Cockcroft-Gault formula or by measure of creatinine clearance from 24 hour urine collection

Other protocol-defined exclusion criteria could apply.

Exclusion Criteria:

* Concurrent treatment with non-permitted drugs and other interventions
* Anticancer treatment within 28 days before the start of trial treatment, for example cyto reductive therapy, radiotherapy (with the exception of palliative bone directed radiotherapy), immune therapy, or cytokine therapy
* Major surgery within 28 days before the start of trial treatment (excluding prior diagnostic biopsy)
* Systemic therapy with immunosuppressive agents within 7 days before the start of trial treatment; or use of any investigational drug within 28 days before the start of trial treatment
* Previous malignant disease other than the target malignancy to be investigated in this trial with the exception of cervical carcinoma in situ and superficial or non invasive bladder cancer (treated with curative intent) within the last 5 years or basal cell or squamous cell carcinoma in situ within the last 3 years
* Rapidly progressive disease which, in the opinion of the Investigator, may predispose to inability to tolerate treatment or trial procedures
* Active or history of central nervous system metastases, except as in the melanoma-specific Central nervous system (CNS) criteria listed above
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that do not require immunosuppression (eg, corneal transplant, hair transplant)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (18):
- Japan (11):
  - NHO Kyushu Cancer Center, Fukuoka
  - National Cancer Center East, Department of Experimental Therapeutics, Kashiwa
  - National Cancer Center East, Department of hepatobiliary and pancreatic oncology, Kashiwa
  - Saitama Cancer Center, Kitaadachi-gun
  - NHO Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center Hospital, Nagoya
  - Kinki University Hospital, Sayama
  - National Cancer Center, Department of Experimental Therapeutics, Tokyo
  - National Cancer Center, Department of hepatobiliary and pancreatic oncology, Tokyo
  - Kanagawa Cancer Center, Department of Gastroenterology, Yokohama
  - Kanagawa Cancer Center, Department of Gastrointestinal Surgery, Yokohama
- South Korea (3):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital; Linkou, Taoyuan District

REFERENCES:
- [Result] Lin CC, Doi T, Muro K, Hou MM, Esaki T, Hara H, Chung HC, Helwig C, Dussault I, Osada M, Kondo S. Bintrafusp Alfa, a Bifunctional Fusion Protein Targeting TGFbeta and PD-L1, in Patients with Esophageal Squamous Cell Carcinoma: Results from a Phase 1 Cohort in Asia. Target Oncol. 2021 Jul;16(4):447-459. doi: 10.1007/s11523-021-00810-9. Epub 2021 Apr 11. PMID 33840050
- [Result] Yoo C, Oh DY, Choi HJ, Kudo M, Ueno M, Kondo S, Chen LT, Osada M, Helwig C, Dussault I, Ikeda M. Phase I study of bintrafusp alfa, a bifunctional fusion protein targeting TGF-beta and PD-L1, in patients with pretreated biliary tract cancer. J Immunother Cancer. 2020 May;8(1):e000564. doi: 10.1136/jitc-2020-000564. PMID 32461347
- [Derived] Vugmeyster Y, Grisic AM, Wilkins JJ, Loos AH, Hallwachs R, Osada M, Venkatakrishnan K, Khandelwal A. Model-informed approach for risk management of bleeding toxicities for bintrafusp alfa, a bifunctional fusion protein targeting TGF-beta and PD-L1. Cancer Chemother Pharmacol. 2022 Oct;90(4):369-379. doi: 10.1007/s00280-022-04468-6. Epub 2022 Sep 6. PMID 36066618
- [Derived] Wilkins JJ, Vugmeyster Y, Dussault I, Girard P, Khandelwal A. Population Pharmacokinetic Analysis of Bintrafusp Alfa in Different Cancer Types. Adv Ther. 2019 Sep;36(9):2414-2433. doi: 10.1007/s12325-019-01018-0. Epub 2019 Jul 5. PMID 31278692
- See also: INTR@PID Clinical Trial Program — http://www.intrapidclinicaltrials.com
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=200647-0008
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation Cohort: M7824 (3 mg/kg): Participants with metastatic or locally advanced solid tumors received intravenous (IV) infusion of M7824 at a dose of 3.0 milligrams per kilogram (mg/kg) over 1 hour once every two weeks for up to 12 months until confirmed progressive disease (PD), unacceptable toxicity, or any criterion for withdrawal from the study or investigational medicinal product (IMP) whichever occurs first.
- Dose Escalation Cohort: M7824 (10 mg/kg): Participants with metastatic or locally advanced solid tumors received intravenous infusion of M7824 at a dose of 10 mg/kg over 1 hour once every two weeks for up to 12 months until confirmed PD, unacceptable toxicity, or any criterion for withdrawal from study or IMP whichever occurs first.
- Dose Escalation Cohort: M7824 (20 mg/kg): Participants with metastatic or locally advanced solid tumors received intravenous infusion of M7824 at a dose of 20 mg/kg over 1 hour once every two weeks for up to 12 months until confirmed PD, unacceptable toxicity, or any criterion for withdrawal from the study or IMP whichever occurs first.
- Expansion Cohort: Biliary Tract Cancer; Expansion Cohort: Gastric Cancer (GC); Expansion Cohort: Esophageal Squamous Cell Cancer: Participants received intravenous infusion of M7824 at a flat dose of 1200 over 1 hour once every two weeks until PD has been confirmed by a subsequent scan, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study or the IMP occurs.
- Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg): Participants received intravenous infusion of M7824 at a dose of 3 mg/kg over 1 hour once every two weeks until PD has been confirmed by a subsequent scan, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study or the IMP occurs.
- Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg): Participants received intravenous infusion of M7824 at a dose of 10 mg/kg over 1 hour once every two weeks until PD has been confirmed by a subsequent scan, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study or the IMP occurs.
Period: Overall Study
Arm/Group | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Dose Escalation Cohort: M7824 (20 mg/kg) | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg)
Started | 4 | 3 | 7 | 30 | 31 | 30 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 4 | 3 | 7 | 30 | 31 | 29 | 3 | 6
Not completed — Death | 3 | 3 | 3 | 23 | 22 | 23 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 5 | 3 | 0 | 1
Not completed — Other | 1 | 0 | 1 | 6 | 4 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Expansion Cohort: Biliary Tract Cancer | Dose Escalation Cohort: M7824 (20 mg/kg) | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg) | Total
Number analyzed (Participants) | 4 | 3 | 30 | 7 | 31 | 30 | 3 | 6 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (8.7) | 57 (18.5) | 63 (9.3) | 54 (10.9) | 62 (11.5) | 60 (9.9) | 58 (16.5) | 56 (13.2) | 61 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 11 | 5 | 5 | 4 | 1 | 1 | 32
  Male | 2 | 0 | 19 | 2 | 26 | 26 | 2 | 5 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity-Japanese | 4 | 3 | 12 | 7 | 12 | 17 | 3 | 6 | 64
  Ethnicity-Korean | 0 | 0 | 15 | 0 | 14 | 3 | 0 | 0 | 32
  Ethnicity-Taiwanese | 0 | 0 | 3 | 0 | 5 | 10 | 0 | 0 | 18
  Race-Asian | 4 | 3 | 30 | 7 | 31 | 30 | 3 | 6 | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: A DLT was defined as any grade greater than or equal to (>=) 3 adverse event suspected to be related to investigational medicinal product (IMP) by the Investigator and / or Sponsor occurring in the DLT evaluation period confirmed by the Safety Monitoring Committee (SMC) to be relevant for the IMP treatment.
Time Frame: Baseline up to Week 3
Population: DLT analysis set included all participants with data used for implementing the dose-escalation schedule. These participants received all study treatment administrations in the DLT evaluation period or stopped treatment because of DLTs in the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Dose Escalation Cohort: M7824 (20 mg/kg)
Number analyzed (Participants) | 4 | 3 | 6
Participants | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) According to National Cancer Institute-Common Terminology Criteria for Adverse Event (NCI-CTCAE) Version 4.03
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs.
Time Frame: First study drug administration up to 30 days after the last drug administration assessed up to approximately 5 years
Population: Safety Analysis Set (SAF) included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Dose Escalation Cohort: M7824 (20 mg/kg) | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg)
Number analyzed (Participants) | 4 | 3 | 7 | 30 | 31 | 30 | 3 | 6
Participants | 4 | 3 | 6 | 28 | 30 | 30 | 2 | 6

3. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (TRAEs) According to NCI-CTCAE Version 4.03
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event needed not necessarily have a causal relationship with the treatment or usage. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: AE with onset after start of treatment or with onset date before the treatment start date but worsening after the treatment start date. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs: reasonably related to the study intervention. Number of participants with TEAEs and treatment related TEAEs were reported.
Time Frame: First study drug administration up to 30 days after the last drug administration assessed up to approximately 5 years
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Dose Escalation Cohort: M7824 (20 mg/kg) | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg)
Number analyzed (Participants) | 4 | 3 | 7 | 30 | 31 | 30 | 3 | 6
Participants | 1 | 2 | 3 | 19 | 16 | 19 | 0 | 0

4. Secondary Outcome: Dose-Escalation Phase: Maximum Serum Concentration (Cmax) of M7824
Description: Cmax is the maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0, 4 hour post dose on Day 1, 2,8,15,29,43
Population: Pharmacokinetic analysis set included all participants who completed at least 1 infusion of M7824, and who provided at least 1 post dose sample with a measurable concentration of M7824. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (mcg/mL)
Groups:
- Pooled Escalation (M7824 3 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [3 mg/kg]): Participants with metastatic or locally advanced solid tumors received intravenous (IV) infusion of M7824 at a dose of 3.0 milligrams per kilogram (mg/kg) over 1 hour once every two weeks for up to 12 months until confirmed progressive disease (PD), unacceptable toxicity, or any criterion for withdrawal from the study or investigational medicinal product (IMP) whichever occurs first in Escalation Cohort or until PD has been confirmed by a subsequent scan, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study or the IMP occurs in Expansion Cohort.
- Pooled Escalation (M7824 10 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [10 mg/kg]): Participants with metastatic or locally advanced solid tumors received intravenous (IV) infusion of M7824 at a dose of 10.0 milligrams per kilogram (mg/kg) over 1 hour once every two weeks for up to 12 months until confirmed progressive disease (PD), unacceptable toxicity, or any criterion for withdrawal from the study or investigational medicinal product (IMP) whichever occurs first in Escalation Cohort or until PD has been confirmed by a subsequent scan, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study or the IMP occurs in Expansion Cohort.
Arm/Group | Pooled Escalation (M7824 3 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [3 mg/kg]) | Pooled Escalation (M7824 10 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [10 mg/kg]) | Dose Escalation Cohort: M7824 (20 mg/kg)
Number analyzed (Participants) | 7 | 9 | 7
Micrograms per milliliter (mcg/mL) | 54.6 (17.9) | 211 (21.7) | 331 (19.2)

5. Secondary Outcome: Dose-Escalation Phase: Terminal Half Life (t1/2) of M7824
Description: t1/2 was the time measured for the concentration to decrease by one half, determined as 0.693/Lambda z, here Lambda z was the terminal elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: Pre-dose, 0, 4 hour post dose on Day 1, 2,8,15,29,43
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Pooled Escalation (M7824 3 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [3 mg/kg]) | Pooled Escalation (M7824 10 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [10 mg/kg]) | Dose Escalation Cohort: M7824 (20 mg/kg)
Number analyzed (Participants) | 4 | 7 | 5
hours | 132 (12.8) | 138 (17.4) | 150 (24.4)

6. Secondary Outcome: Dose-Escalation Phase: Area Under the Serum Concentration Time Curve From Zero to Last Sampling Time (AUC0-t) of M7824
Description: Area under the serum concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated by linear trapezoidal summation.
Time Frame: Pre-dose, 0, 4 hour post dose on Day 1, 2, 8, 15, 29, 43
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter(hr*mcg/mL)
Arm/Group | Pooled Escalation (M7824 3 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [3 mg/kg]) | Pooled Escalation (M7824 10 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [10 mg/kg]) | Dose Escalation Cohort: M7824 (20 mg/kg)
Number analyzed (Participants) | 7 | 8 | 6
hour*microgram per milliliter(hr*mcg/mL) | 7940 (16.7) | 29200 (25.3) | 51300 (24.7)

7. Secondary Outcome: Dose-Escalation Phase: Area Under The Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of M7824
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: Pre-dose, 0, 4 hour post dose on Day 1, 2, 8, 15, 29, 43
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mcg/mL
Arm/Group | Pooled Escalation (M7824 3 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [3 mg/kg]) | Pooled Escalation (M7824 10 mg/kg) and Expansion Cohort (Hepatocellular Carcinoma [10 mg/kg]) | Dose Escalation Cohort: M7824 (20 mg/kg)
Number analyzed (Participants) | 7 | 7 | 5
hr*mcg/mL | 9600 (15.2) | 34600 (29.7) | 61700 (26.6)

8. Secondary Outcome: Dose-Escalation Phase: Number of Participants With Positive Serum Titers of Anti-Drug Antibodies of M7824
Description: The detection of antibodies to M7824 was performed using a validated electrochemiluminescence (ECL) immunoassay with tiered testing of screening, confirmatory and titration. Number of participants with positive anti-drug antibody (ADA) of M7824 were reported.
Time Frame: Predose, Day 15, 43, 85 and every 6-weekly until progression or end of the treatment whichever occur first, assessed up to 3 years
Population: Immunogenicity Analysis Set included participants who received at least 1 dose of study drug and who had at least 1 valid result of ADA at any time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Dose Escalation Cohort: M7824 (20 mg/kg)
Number analyzed (Participants) | 4 | 3 | 6
Participants | 1 | 0 | 3

9. Secondary Outcome: Dose-Escalation Part: Number of Participants With Best Overall Response (BOR) As Assessed By Investigator
Description: BOR was assessed by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. BOR was defined as sum of complete response and partial response (CR+PR). For target lesions (TLs), CR was defined as the disappearance of all TLs; PR was defined as at least a 30 percent (%) decrease in the sum of largest diameter (SLD) of the TLs, taking as a reference the baseline SLD.
Time Frame: Date of randomization up to 2 years
Population: Full analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Dose Escalation Cohort: M7824 (20 mg/kg)
Number analyzed (Participants) | 4 | 3 | 7
Participants
  Complete response | 0 | 0 | 0
  Partial response | 1 | 0 | 1
  Stable disease | 2 | 1 | 0
  Progressive disease | 1 | 2 | 4
  Not evaluable | 0 | 0 | 2

10. Secondary Outcome: Expansion Part: Best Overall Response (BOR) As Assessed By Investigator
Description: BOR was assessed by investigator according to RECIST Version 1.1. BOR was defined as sum of CR and PR. For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30 percent (%) decrease in the SLD of the TLs, taking as a reference the baseline SLD.
Time Frame: Date of randomization up to 2 years
Population: Full analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer
Number analyzed (Participants) | 30 | 31 | 30
Participants
  Complete response | 1 | 2 | 0
  Partial response | 6 | 5 | 6
  Stable disease | 4 | 5 | 5
  Progressive disease | 17 | 16 | 17
  Not evaluable | 2 | 3 | 2

11. Secondary Outcome: Expansion Part: BOR According to RECIST 1.1 As Adjudicated By The Independent Review Committee (IRC)
Description: The BOR per Independent Endpoint Review Committee (IRC) adjudication was determined according to RECIST 1.1. BOR is defined as sum of CR and PR. For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30 percent (%) decrease in the SLD of the TLs, taking as a reference the baseline SLD.
Time Frame: Up to 2 years
Population: Full analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg): Participants with HCC received intravenous infusion of M7824 at a dose of 3 mg/kg over 1 hour once every two weeks until PD has been confirmed by a subsequent scan, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study or the IMP occurs.
Arm/Group | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg)
Number analyzed (Participants) | 30 | 31 | 30 | 3 | 6
Participants
  Complete response (CR) | 2 | 3 | 0 | 0 | 0
  Partial Response (PR) | 4 | 3 | 3 | 0 | 0
  Stable disease (SD) | 6 | 2 | 3 | 1 | 0
  Non-CR/Non-PD | 0 | 0 | 3 | 0 | 0
  Progressive disease (PD) | 16 | 21 | 18 | 1 | 6
  Not evaluable (NE) | 2 | 2 | 3 | 1 | 0

12. Secondary Outcome: Expansion Part: Duration of Response (DOR)
Description: Duration of response according to RECIST 1.1 as adjudicated by the IRC was defined as the time from first confirmed response until the first documented disease progression that was subsequently confirmed. It was analyzed using Kaplan-Meier method.
Time Frame: Up to 2 years
Population: Full analysis set included all participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer
Number analyzed (Participants) | 30 | 31 | 30
Months | NA [8.3 to 34.5] — Due to small number of events, Median from Kaplan-Meier survival curves could not derive. | 20.8 [2.4 to 29.0] | 7.0 [2.8 to 24.9]

13. Secondary Outcome: Expansion Part: Disease Control Rate
Description: The disease control rate was defined as the percentage of participants with BOR. The BOR per IRC adjudication was determined according to RECIST 1.1. BOR is defined as sum of CR and PR. For TLs, CR was defined as the disappearance of all TLs; PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline SLD.
Time Frame: Up to 2 years
Population: Full analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Expansion Cohort: Hepatocellular Carcinoma (3mg/kg): Participants with HCC received intravenous infusion of M7824 at a dose of 3 mg/kg over 1 hour once every two weeks until PD has been confirmed by a subsequent scan, unacceptable toxicity, or occurrence of any criterion for withdrawal from the study or the IMP occurs.
Arm/Group | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg)
Number analyzed (Participants) | 30 | 31 | 30 | 3 | 6
Percentage of Participants | 40.0 [22.7 to 59.4] | 22.6 [11.9 to 44.6] | 20 [14.7 to 49.4] | 1 [0.8 to 90.6] | 0 [0.0 to 45.9]

14. Secondary Outcome: Expansion Part: Progression Free Survival (PFS) Time
Description: PFS was defined as the time from date of randomization until date of the first documentation of progressive disease (PD) or death due to any cause in the absence of documented PD, whichever occurs first. PFS was assessed as RECIST v1.1 as adjudicated by IRC. PD is defined as at least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Date of randomization until death or progressive disease assessed up to 2 years
Population: Full analysis set included all participants who received at least 1 dose of study treatment. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg)
Number analyzed (Participants) | 25 | 25 | 26 | 3 | 6
Months | 2.5 [0.0 to 38.6] | 1.3 [0.4 to 31.6] | 1.4 [0.0 to 30.3] | 2.1 [1.3 to 2.8] | 1.2 [0.8 to 2.7]

15. Secondary Outcome: Expansion Part: Overall Survival (OS) Time
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Date of randomization until death assessed up to 2 years
Population: Full analysis set included all participants who received at least 1 dose of study treatment. "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg)
Number analyzed (Participants) | 19 | 21 | 6 | 3 | 6
Months | 12.7 [1.9 to 38.7] | 10.1 [0.5 to 38.3] | 11.9 [0.1 to 38.0] | 4.4 [4.3 to 6.9] | 4.0 [2.1 to NA] — Due to small number of events, Upper limit from Kaplan-Meier survival curves could not derive.

ADVERSE EVENTS:
Time Frame: First study drug administration up to 30 days after the last drug administration assessed up to approximately up to 5 years.
Arm/Group | Expansion Cohort: Biliary Tract Cancer | Expansion Cohort: Gastric Cancer (GC) | Expansion Cohort: Esophageal Squamous Cell Cancer | Dose Escalation Cohort: M7824 (3 mg/kg) | Dose Escalation Cohort: M7824 (10 mg/kg) | Dose Escalation Cohort: M7824 (20 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg)
All-Cause Mortality (participants affected / at risk) | 23/30 | 22/31 | 24/30 | 3/4 | 3/3 | 3/7 | 3/3 | 5/6
Serious Adverse Events (participants affected / at risk) | 18/30 | 18/31 | 14/30 | 4/4 | 0/3 | 5/7 | 2/3 | 3/6
Other Adverse Events (participants affected / at risk) | 28/30 | 30/31 | 30/30 | 4/4 | 3/3 | 6/7 | 1/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expansion Cohort: Biliary Tract Cancer (N=30) | Expansion Cohort: Gastric Cancer (GC) (N=31) | Expansion Cohort: Esophageal Squamous Cell Cancer (N=30) | Dose Escalation Cohort: M7824 (3 mg/kg) (N=4) | Dose Escalation Cohort: M7824 (10 mg/kg) (N=3) | Dose Escalation Cohort: M7824 (20 mg/kg) (N=7) | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) (N=3) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg) (N=6)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kaposi's varicelliform eruption (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expansion Cohort: Biliary Tract Cancer (N=30) | Expansion Cohort: Gastric Cancer (GC) (N=31) | Expansion Cohort: Esophageal Squamous Cell Cancer (N=30) | Dose Escalation Cohort: M7824 (3 mg/kg) (N=4) | Dose Escalation Cohort: M7824 (10 mg/kg) (N=3) | Dose Escalation Cohort: M7824 (20 mg/kg) (N=7) | Expansion Cohort: Hepatocellular Carcinoma (3 mg/kg) (N=3) | Expansion Cohort: Hepatocellular Carcinoma (10 mg/kg) (N=6)
Anaemia (Blood and lymphatic system disorders) | 10 (15) | 11 (16) | 7 (11) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epidermal naevus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vasculitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 6 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 7 (7) | 5 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (5) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal mucosal hyperplasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 6 (7) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (5) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 13 (22) | 7 (10) | 5 (5) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis chronic active (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pitted keratolysis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 7 (8) | 4 (4) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (7) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Zinc deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (4) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (8) | 1 (9) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 7 (7) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (6) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (8) | 7 (9) | 6 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fibrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data collection and analysis of Pharmacokinetics of Cmin was omitted and not conducted due to business reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02699515/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT02699515/SAP_001.pdf